CLINICAL TRIAL: NCT01938430
Title: A Phase 2, Multicenter, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Ledipasvir Fixed-Dose Combination + Ribavirin Administered in Subjects Infected With Chronic HCV Who Have Advanced Liver Disease or Are Post-Liver Transplant
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination + Ribavirin in Subjects With Chronic HCV With Advanced Liver Disease or Post-Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0123
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-03

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Cohort A, Group 1 (12 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 1 (24 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 2 (12 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 2 (24 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3.
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with Fibrosis Stage F0-F3
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 4 (12 wk): CPT Class A (5-6) (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with CPT Class A (CPT score 5-6)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 4 (24 wk): CPT Class A (5-6) (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with CPT Class A (CPT score 5-6)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 5 (12 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 5 (24 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 6 (12 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 6 (24 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 7 (12 wk): FCH (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with FCH
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 7 (24 wk): FCH (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with FCH
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — RBV tablets administered orally in a divided daily dose

SUMMARY:
This study will evaluate ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) plus ribavirin (RBV) in participants with advanced liver disease or posttransplant and chronic genotype 1 or 4 hepatitis C virus (HCV) infection.

* Cohort A: decompensated cirrhosis (advanced liver disease), no prior liver transplant;
* Cohort B: post-liver transplant, with or without cirrhosis;
* Group assignment within cohorts is based on severity of liver impairment at screening (Child-Pugh-Turcotte (CPT) score for participants with cirrhosis; fibrosis; or presence of disease for fibrosing cholestatic hepatitis (FCH) groups)
* Randomization is 1:1 within groups to 12 or 24 weeks of LDV/SOF+RBV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Chronic genotype 1 or 4 HCV infection
* Normal ECG
* Negative serum pregnancy test for female subjects
* Male subjects and female subjects of childbearing potential must agree to use contraception
* Able to comply with the dosing instructions for study drug and able to complete the study schedule of assessments, including all required post treatment visits

Exclusion Criteria:

* Serious or active medical or psychiatric illness
* HIV or hepatitis B viral (HBV) infection
* Stomach disorder that could interfere with the absorption of the study drug
* Treated with an anti-HCV medication in the last 30 days
* Any prior exposure to an HCV nonstructural protein (NS)5a-specific inhibitor
* Use of human granulocyte-macrophage colony-stimulating factor (GM-CSF), epoetin alfa or other therapeutic hematopoietic agents within 2 weeks of screening
* History of clinically significant medical condition associated with other chronic liver disease
* Active spontaneous bacterial peritonitis at screening
* Females who are breastfeeding
* Infection requiring systemic antibiotics
* Participated in a clinical study with an investigational drug or biologic within the last 30 days
* Active or history (last 6 months) of drug or alcohol abuse
* History of organ transplant other than liver or kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shampa De-Oertel, PhD, Study Director — Gilead Sciences
Locations (28):
- United States (28):
  - Phoenix, Arizona
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Murray, Utah
  - Richmond, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Welzel TM, Reddy KR, Flamm SL, Denning J, Lin M, Hyland R, Pang PS, McHutchison JG, Charlton M, Everson GT, Zeuzem S, Afdhal N. On-treatment HCV RNA in patients with varying degrees of fibrosis and cirrhosis in the SOLAR-1 trial. Antivir Ther. 2016;21(6):541-546. doi: 10.3851/IMP3037. Epub 2016 Feb 18. PMID 26891418
- [Derived] Charlton M, Everson GT, Flamm SL, Kumar P, Landis C, Brown RS Jr, Fried MW, Terrault NA, O'Leary JG, Vargas HE, Kuo A, Schiff E, Sulkowski MS, Gilroy R, Watt KD, Brown K, Kwo P, Pungpapong S, Korenblat KM, Muir AJ, Teperman L, Fontana RJ, Denning J, Arterburn S, Dvory-Sobol H, Brandt-Sarif T, Pang PS, McHutchison JG, Reddy KR, Afdhal N; SOLAR-1 Investigators. Ledipasvir and Sofosbuvir Plus Ribavirin for Treatment of HCV Infection in Patients With Advanced Liver Disease. Gastroenterology. 2015 Sep;149(3):649-59. doi: 10.1053/j.gastro.2015.05.010. Epub 2015 May 15. PMID 25985734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 06 September 2013. The last study visit occurred on 25 March 2015.
Pre-assignment Details: * Cohort A: decompensated cirrhosis (advanced liver disease), no prior liver transplant;
  * Cohort B: post-liver transplant, with or without cirrhosis;
  * Group assignment within cohorts was based on severity of liver impairment at screening (or presence of disease for FCH groups);
  * Randomization was 1:1 within groups to 12 or 24 weeks of treatment.
Groups:
- Cohort A, Group 1 (12 wk): CPT Class B (7-9): Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily plus ribavirin (RBV) tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with Child-Pugh-Turcotte (CPT) Class B (CPT score 7-9).
  CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15 (maximum score for study was 12); higher scores indicate greater severity of disease.
- Cohort A, Group 1 (24 wk): CPT Class B (7-9); Cohort B, Group 5 (24 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9)
- Cohort A, Group 2 (12 wk): CPT Class C (10-12); Cohort B, Group 6 (12 wk): CPT Class C (10-12): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12)
- Cohort A, Group 2 (24 wk): CPT Class C (10-12); Cohort B, Group 6 (24 wk): CPT Class C (10-12): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12)
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3
  F0: no fibrosis; F1: portal fibrosis without septa; F2: portal fibrosis with rare septa, F3: numerous septa without cirrhosis; F4: cirrhosis
- Cohort B, Group 3 (24 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with Fibrosis Stage F0-F3
- Cohort B, Group 4 (12 wk): CPT Class A (5-6): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with CPT Class A (CPT score 5-6)
- Cohort B, Group 4 (24 wk): CPT Class A (5-6): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with CPT Class A (CPT score 5-6)
- Cohort B, Group 5 (12 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
- Cohort B, Group 7 (12 wk): FCH: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with fibrosing cholestatic hepatitis (FCH)
- Cohort B, Group 7 (24 wk): FCH: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with FCH
Period: Overall Study
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Started | 30 | 29 | 23 | 26 | 55 | 56 | 26 | 25 | 26 | 26 | 6 | 4 | 4 | 3
Completed | 26 | 26 | 18 | 24 | 55 | 55 | 24 | 24 | 22 | 23 | 3 | 3 | 4 | 2
Not Completed | 4 | 3 | 5 | 2 | 0 | 1 | 2 | 1 | 4 | 3 | 3 | 1 | 0 | 1
Not completed — Randomized but Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least one dose of study drug
Groups:
- Cohort A, Group 1 (12 wk): CPT Class B (7-9); Cohort B, Group 5 (12 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3
- Total: Total of all reporting groups
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH | Total
Number analyzed (Participants) | 30 | 29 | 23 | 26 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.1) | 58 (6.5) | 57 (6.2) | 59 (4.6) | 59 (6.6) | 58 (6.4) | 61 (6.2) | 61 (10.4) | 59 (5.8) | 61 (6.6) | 60 (3.8) | 61 (1.7) | 62 (3.2) | 58 (8.5) | 59 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 9 | 8 | 10 | 10 | 7 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 73
  Male | 22 | 18 | 14 | 18 | 45 | 46 | 19 | 22 | 22 | 23 | 5 | 4 | 4 | 2 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 2 | 4 | 4 | 6 | 2 | 2 | 5 | 3 | 3 | 0 | 0 | 0 | 38
  Not Hispanic or Latino | 26 | 26 | 21 | 22 | 51 | 50 | 24 | 23 | 21 | 23 | 2 | 4 | 4 | 2 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 3 | 2 | 1 | 4 | 4 | 3 | 4 | 5 | 2 | 1 | 0 | 0 | 0 | 30
  White | 29 | 26 | 21 | 24 | 50 | 49 | 21 | 20 | 21 | 24 | 4 | 4 | 4 | 2 | 299
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 23 | 26 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2 | 337
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.68) | 5.8 (0.82) | 5.6 (0.62) | 5.8 (0.71) | 6.5 (0.62) | 6.4 (0.93) | 6.2 (0.77) | 6.7 (0.34) | 6.3 (0.55) | 6.2 (0.67) | 6.4 (0.42) | 6.3 (0.37) | 6.5 (1.24) | 7.1 (0.90) | 6.2 (0.77)
HCV RNA Category [Number; unit: participants]
  < 800 IU/mL | 14 | 11 | 14 | 15 | 10 | 10 | 7 | 0 | 6 | 9 | 1 | 0 | 1 | 0 | 98
  ≥ 800 IU/mL | 16 | 18 | 9 | 11 | 45 | 46 | 19 | 25 | 20 | 17 | 4 | 4 | 3 | 2 | 239
HCV Genotype [Number; unit: participants]
  Genotype 1a | 19 | 22 | 15 | 18 | 40 | 40 | 17 | 17 | 20 | 18 | 4 | 3 | 3 | 2 | 238
  Genotype 1b | 10 | 7 | 6 | 8 | 14 | 16 | 9 | 8 | 6 | 7 | 1 | 1 | 1 | 0 | 94
  Genotype 4 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 5 | 6 | 7 | 11 | 10 | 7 | 1 | 3 | 5 | 2 | 1 | 0 | 0 | 62
    CT | 20 | 18 | 13 | 15 | 33 | 27 | 11 | 19 | 14 | 16 | 2 | 2 | 2 | 1 | 193
    TT | 6 | 6 | 4 | 4 | 11 | 19 | 8 | 5 | 9 | 5 | 1 | 1 | 2 | 1 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 12 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 22 | 23 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 86.7 | 88.9 | 86.4 | 87.0 | 96.4 | 98.2 | 96.2 | 96.0 | 84.6 | 88.5 | 60.0 | 75.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 26 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants
  Discontinued LDV/SOF | 0.0 | 6.9 | 4.3 | 7.7 | 0.0 | 3.6 | 3.8 | 0.0 | 7.7 | 11.5 | 0.0 | 0.0 | 0.0 | 0.0
  Discontinued Any Study Drug | 0.0 | 13.8 | 13.0 | 34.6 | 10.9 | 17.9 | 15.4 | 8.0 | 23.1 | 34.6 | 40.0 | 25.0 | 25.0 | 0.0

3. Secondary Outcome: Percentage of Participants With SVR 2 Weeks After Discontinuation of Therapy (SVR2)
Description: SVR2 was defined as HCV RNA < LLOQ at 2 weeks after stopping study treatment.
Time Frame: Posttreatment Week 2
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 2 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 22 | 24 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 96.7 | 92.6 | 95.5 | 95.8 | 100.0 | 98.2 | 96.2 | 100.0 | 88.5 | 92.3 | 100.0 | 75.0 | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants With SVR 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 4 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 22 | 23 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 90.0 | 88.9 | 90.9 | 95.7 | 96.4 | 98.2 | 96.2 | 100.0 | 88.5 | 92.3 | 100.0 | 75.0 | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants With SVR 8 Weeks After Discontinuation of Therapy (SVR8)
Description: SVR8 was defined as HCV RNA < LLOQ at 8 weeks after stopping study treatment.
Time Frame: Posttreatment Week 8
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 8 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 22 | 23 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 86.7 | 88.9 | 86.4 | 95.7 | 96.4 | 98.2 | 96.2 | 100.0 | 88.5 | 88.5 | 60.0 | 75.0 | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants With SVR 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 24 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 21 | 23 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 86.7 | 88.9 | 85.7 | 87.0 | 96.4 | 98.2 | 96.2 | 96.0 | 84.6 | 88.5 | 60.0 | 75.0 | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ on 2 consecutive measurements while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set. Participants were excluded from the analysis if they received a liver transplant while on study (with HCV RNA <LLOQ at transplant) prior to lower bound of Posttreatment Week 12 visit window.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 22 | 23 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 10.0 | 3.7 | 4.5 | 8.7 | 3.6 | 0.0 | 0.0 | 0.0 | 3.8 | 0.0 | 40.0 | 25.0 | 3.6 | 0.0

8. Secondary Outcome: Percentage of Participants With Posttransplant Virologic Response (pTVR) at Posttransplant Week 12
Description: pTVR was defined as HCV RNA < LLOQ at Week 12 after transplant.
Time Frame: Posttransplant Week 12
Population: Participants who had a liver transplant while on study were analyzed if their last observed HCV RNA measurement prior to transplant was < LLOQ. Participants who received a transplant from an HCV-infected donor were excluded from analysis.
Measure: Number; unit: percentage of participants
Groups:
- All LDV/SOF+RBV: All participants in the analysis are presented in a single group, regardless of randomization group assignment.
Arm/Group | All LDV/SOF+RBV
Number analyzed (Participants) | 7
percentage of participants | 85.7

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 26 | 55 | 56 | 26 | 25 | 26 | 26 | 5 | 4 | 4 | 2
percentage of participants | 6.7 | 6.9 | 13.0 | 3.8 | 16.4 | 12.5 | 15.4 | 4.0 | 3.8 | 7.7 | 0.0 | 0.0 | 25.0 | 0.0

10. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 26 | 55 | 55 | 26 | 25 | 25 | 26 | 5 | 4 | 4 | 2
percentage of participants | 36.7 | 41.4 | 39.1 | 38.5 | 49.1 | 41.8 | 34.6 | 28.0 | 8.0 | 42.3 | 40.0 | 25.0 | 50.0 | 0.0

11. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 26 | 55 | 55 | 26 | 25 | 25 | 26 | 5 | 4 | 4 | 2
percentage of participants | 83.3 | 82.8 | 100.0 | 84.6 | 87.3 | 90.9 | 88.5 | 80.0 | 72.0 | 88.5 | 100.0 | 100.0 | 100.0 | 50.0

12. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 6
Time Frame: Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 22 | 26 | 55 | 55 | 25 | 25 | 25 | 26 | 5 | 4 | 4 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 96.2 | 96.4 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 50.0

13. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 22 | 25 | 55 | 55 | 25 | 25 | 25 | 26 | 5 | 4 | 4 | 2
percentage of participants | 100.0 | 96.6 | 100.0 | 92.0 | 100.0 | 100.0 | 100.0 | 100.0 | 96.0 | 96.2 | 100.0 | 100.0 | 100.0 | 50.0

14. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 21 | 24 | 55 | 54 | 25 | 25 | 23 | 25 | 5 | 4 | 4 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 96.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

15. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 16
Time Frame: Week 16
Population: Participants in the Full Analysis Set who were randomized to a 24-week treatment group and had available data were analyzed. 12-week treatment groups (did not collect data past Week 12) are not presented in this table.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 27 | 22 | 54 | 25 | 22 | 4 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

16. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 20
Time Frame: Week 20
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 27 | 22 | 54 | 25 | 22 | 4 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

17. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 24
Time Frame: Week 24
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 22 | 51 | 25 | 22 | 3 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

18. Secondary Outcome: HCV RNA and Change From Baseline at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 24 | 55 | 55 | 25 | 24 | 25 | 26 | 4 | 4 | 4 | 2
log10 IU/mL
  Week 1 | 2.26 (0.695) | 2.49 (0.830) | 2.11 (0.643) | 2.46 (0.968) | 2.33 (0.983) | 2.42 (0.730) | 2.40 (0.890) | 2.86 (0.792) | 2.84 (0.678) | 2.56 (0.774) | 2.76 (0.571) | 2.75 (1.065) | 2.28 (1.149) | 4.30 (1.424)
  Change at Week 1 | -3.59 (0.476) | -3.34 (0.658) | -3.47 (0.579) | -3.32 (0.669) | -4.14 (0.721) | -3.98 (0.682) | -3.80 (0.712) | -3.86 (0.759) | -3.41 (0.409) | -3.68 (0.506) | -3.75 (0.584) | -3.52 (1.028) | -4.22 (0.864) | -2.76 (0.526)

19. Secondary Outcome: HCV RNA and Change From Baseline at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 24 | 54 | 52 | 25 | 25 | 25 | 26 | 5 | 4 | 4 | 1
log10 IU/mL
  Week 2 | 1.60 (0.484) | 1.67 (0.574) | 1.49 (0.404) | 1.82 (0.748) | 1.64 (0.751) | 1.59 (0.516) | 1.73 (0.631) | 1.91 (0.641) | 2.03 (0.585) | 1.76 (0.628) | 1.80 (0.645) | 2.00 (0.746) | 1.66 (0.637) | 1.61 (NA) — 1 participant analyzed: SD not calculable
  Change at Week 2 | -4.25 (0.575) | -4.16 (0.748) | -4.09 (0.604) | -3.98 (0.581) | -4.83 (0.720) | -4.79 (0.845) | -4.48 (0.668) | -4.84 (0.636) | -4.22 (0.489) | -4.47 (0.503) | -4.56 (0.765) | -4.26 (0.825) | -4.85 (1.090) | -4.81 (NA) — 1 participant analyzed: standard deviation (SD) not calculable

20. Secondary Outcome: HCV RNA and Change From Baseline at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 23 | 25 | 55 | 55 | 26 | 25 | 25 | 26 | 5 | 4 | 4 | 2
log10 IU/mL
  Week 4 | 1.20 (0.117) | 1.21 (0.153) | 1.15 (0.000) | 1.23 (0.265) | 1.24 (0.271) | 1.16 (0.065) | 1.18 (0.120) | 1.23 (0.212) | 1.24 (0.184) | 1.18 (0.150) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.67 (0.738)
  Change at Week 4 | -4.65 (0.668) | -4.63 (0.789) | -4.44 (0.618) | -4.56 (0.655) | -5.23 (0.629) | -5.24 (0.929) | -5.01 (0.736) | -5.52 (0.376) | -5.01 (0.537) | -5.05 (0.662) | -5.21 (0.422) | -5.12 (0.368) | -5.36 (1.237) | -5.39 (0.159)

21. Secondary Outcome: HCV RNA and Change From Baseline at Week 6
Time Frame: Baseline; Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 29 | 22 | 26 | 54 | 55 | 25 | 25 | 25 | 26 | 5 | 4 | 4 | 1
log10 IU/mL
  Week 6 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.042) | 1.15 (0.004) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (NA) — 1 participant analyzed: SD not calculable
  Change at Week 6 | -4.70 (0.676) | -4.69 (0.822) | -4.47 (0.616) | -4.61 (0.695) | -5.32 (0.618) | -5.25 (0.936) | -5.05 (0.788) | -5.60 (0.345) | -5.10 (0.559) | -5.09 (0.669) | -5.21 (0.422) | -5.12 (0.368) | -5.36 (1.237) | -5.28 (NA) — 1 participant analyzed: SD not calculable

22. Secondary Outcome: HCV RNA and Change From Baseline at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 28 | 22 | 24 | 55 | 55 | 25 | 25 | 24 | 25 | 5 | 4 | 4 | 2
log10 IU/mL
  Week 8 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.16 (0.081) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.22 (0.110)
  Change at Week 8 | -4.70 (0.676) | -4.67 (0.834) | -4.47 (0.616) | -4.61 (0.715) | -5.33 (0.615) | -5.25 (0.936) | -5.05 (0.788) | -5.60 (0.345) | -5.11 (0.571) | -5.10 (0.682) | -5.21 (0.422) | -5.12 (0.368) | -5.36 (1.237) | -5.83 (0.787)

23. Secondary Outcome: HCV RNA and Change From Baseline at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 30 | 27 | 21 | 24 | 55 | 54 | 24 | 25 | 23 | 25 | 5 | 4 | 4 | 2
log10 IU/mL
  Week 12 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Change at Week 12 | -4.70 (0.676) | -4.70 (0.842) | -4.44 (0.614) | -4.62 (0.737) | -5.33 (0.615) | -5.25 (0.943) | -5.09 (0.781) | -5.60 (0.345) | -5.14 (0.562) | -5.10 (0.682) | -5.21 (0.422) | -5.12 (0.368) | -5.36 (1.237) | -5.91 (0.897)

24. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 4 in MELD Score
Description: Model for End-Stage Liver Disease (MELD) scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40; higher scores/increased scores indicate greater severity of disease.
Time Frame: Baseline to Posttreatment Week 4
Population: Full Analysis Set. Participants with cirrhosis were analyzed if they had measurements at both baseline and Posttreatment Week 4. Only groups with cirrhotic participants are presented.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12)
Number analyzed (Participants) | 28 | 25 | 21 | 20 | 23 | 25 | 21 | 20 | 5 | 3
percentage of participants
  Decrease | 60.7 | 68.0 | 61.9 | 80.0 | 30.4 | 52.0 | 66.7 | 70.0 | 40.0 | 66.7
  No Change | 17.9 | 20.0 | 9.5 | 15.0 | 39.1 | 16.0 | 19.0 | 5.0 | 20.0 | 0.0
  Increase | 21.4 | 12.0 | 28.6 | 5.0 | 30.4 | 32.0 | 14.3 | 25.0 | 40.0 | 33.3

25. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 4 in CPT Score
Description: CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15 (maximum score for entry into the study was 12); higher scores/increased scores indicate greater severity of disease. Groups are arranged by cohort, then by duration of treatment, then by CPT class at baseline.
Time Frame: Baseline to Posttreatment Week 4
Population: Full Analysis Set. Cirrhotic participants were analyzed if they had measurements at both baseline and Posttreatment Week 4. Only groups with cirrhotic participants are presented.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A: Baseline CPT Class A (24 wk): Includes participants in Cohort A (24 wk) with CPT score A at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class B (12 wk): Includes participants in Cohort A (12 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class B (24 wk): Includes participants in Cohort A (24 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class C (12 wk): Includes participants in Cohort A (12 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class C (24 wk): Includes participants in Cohort A (24 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class A (12 wk): Includes participants in Cohort B (12 wk) with CPT score A at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class A (24 wk): Includes participants in Cohort B (24 wk) with CPT score A at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class B (12 wk): Includes participants in Cohort B (12 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class B (24 wk): Includes participants in Cohort B (24 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class C (12 wk): Includes participants in Cohort B (12 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class C (24 wk): Includes participants in Cohort B (24 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
Arm/Group | Cohort A: Baseline CPT Class A (24 wk) | Cohort A: Baseline CPT Class B (12 wk) | Cohort A: Baseline CPT Class B (24 wk) | Cohort A: Baseline CPT Class C (12 wk) | Cohort A: Baseline CPT Class C (24 wk) | Cohort B: Baseline CPT Class A (12 wk) | Cohort B: Baseline CPT Class A (24 wk) | Cohort B: Baseline CPT Class B (12 wk) | Cohort B: Baseline CPT Class B (24 wk) | Cohort B: Baseline CPT Class C (12 wk) | Cohort B: Baseline CPT Class C (24 wk)
Number analyzed (Participants) | 1 | 30 | 26 | 19 | 18 | 22 | 23 | 23 | 22 | 4 | 3
percentage of participants
  Decrease | 0.0 | 63.3 | 50.0 | 89.5 | 72.2 | 18.2 | 47.8 | 56.5 | 59.1 | 50.0 | 100.0
  No Change | 0.0 | 23.3 | 38.5 | 10.5 | 27.8 | 68.2 | 52.2 | 34.8 | 31.8 | 50.0 | 0.0
  Increase | 100.0 | 13.3 | 11.5 | 0.0 | 0.0 | 13.6 | 0.0 | 8.7 | 9.1 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks on treatment plus 30 days
Description: Safety Analysis Set: participants who were enrolled and received at least one dose of study drug
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Serious Adverse Events (participants affected / at risk) | 3/30 | 10/29 | 6/23 | 11/26 | 6/55 | 12/56 | 3/26 | 4/25 | 5/26 | 11/26 | 1/5 | 3/4 | 1/4 | 1/2
Other Adverse Events (participants affected / at risk) | 26/30 | 28/29 | 22/23 | 26/26 | 54/55 | 54/56 | 25/26 | 23/25 | 23/26 | 26/26 | 5/5 | 4/4 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Group 1 (12 wk): CPT Class B (7-9) (N=30) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) (N=29) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) (N=23) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) (N=26) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (N=55) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (N=56) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) (N=26) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) (N=25) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) (N=26) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) (N=26) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) (N=5) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) (N=4) | Cohort B, Group 7 (12 wk): FCH (N=4) | Cohort B, Group 7 (24 wk): FCH (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complications of transplanted liver (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Group 1 (12 wk): CPT Class B (7-9) (N=30) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) (N=29) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) (N=23) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) (N=26) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (N=55) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (N=56) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) (N=26) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) (N=25) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) (N=26) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) (N=26) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) (N=5) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) (N=4) | Cohort B, Group 7 (12 wk): FCH (N=4) | Cohort B, Group 7 (24 wk): FCH (N=2)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 4 | 11 | 24 | 18 | 8 | 8 | 7 | 10 | 4 | 2 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 2 | 3 | 4 | 5 | 1 | 1 | 2 | 5 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 3 | 2 | 0 | 1 | 3 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 7 | 4 | 4 | 2 | 1 | 4 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 7 | 8 | 8 | 9 | 15 | 2 | 3 | 2 | 5 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 5 | 5 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 11 | 9 | 13 | 10 | 21 | 7 | 5 | 5 | 8 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 5 | 5 | 9 | 3 | 3 | 3 | 8 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 17 | 15 | 13 | 12 | 34 | 31 | 16 | 10 | 12 | 11 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 0 | 7 | 2 | 3 | 1 | 5 | 4 | 4 | 1 | 2 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Pseudocyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2 | 6 | 5 | 5 | 0 | 1 | 2 | 5 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2 | 0 | 6 | 5 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 5 | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 1 | 4 | 9 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 8 | 3 | 5 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 3 | 5 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 4 | 6 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 1 | 3 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 6 | 3 | 7 | 6 | 10 | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 12 | 7 | 5 | 17 | 19 | 7 | 5 | 7 | 9 | 3 | 1 | 2 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 3 | 0 | 3 | 2 | 5 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 7 | 4 | 8 | 8 | 11 | 5 | 3 | 1 | 3 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 4 | 3 | 2 | 3 | 5 | 9 | 3 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4 | 4 | 4 | 5 | 7 | 3 | 0 | 4 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 4 | 13 | 6 | 5 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 5 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 6 | 2 | 1 | 6 | 1 | 4 | 2 | 0 | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 3 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 2 | 7 | 10 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years